CLINICAL TRIAL: NCT03115216
Title: The Femtosecond Laser in Residency Training (FLIRT) Pilot Study: Femtosecond Laser-Assisted Versus Manual Cataract Extraction and Intraocular Lens Implantation
Brief Title: The Femtosecond Laser in Residency Training (FLIRT) Pilot Study
Acronym: FLIRT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn during planning stages
Sponsor: University of Southern California (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLIRT
Record Dates: First submitted 2016-11-15; First posted 2017-04-14 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2017-04

CONDITIONS: Cataract; Intraocular Lens Implantation
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLA-CEIOL (Active Comparator): Femtosecond laser assisted cataract extraction and intraocular lens placement
  Interventions: Procedure: FLA-CEIOL
- CEIOL (Active Comparator): Clear corneal incision with manual cataract extraction and intraocular lens placement
  Interventions: Procedure: CEIOL

INTERVENTIONS:
Procedure: FLA-CEIOL — Femtosecond laser-assisted cataract extraction and intraocular lens placement
  Arms: FLA-CEIOL
Procedure: CEIOL — Manual cataract extraction and intraocular lens placement
  Arms: CEIOL

SUMMARY:
This pilot study aims to primarily assess the rate of complication of anterior vitrectomy for patients undergoing femtosecond laser-assisted (FLA) cataract extraction and intraocular lens placement (CEIOL) compared to manual CEIOL, when performed by resident physicians under direct attending supervision. In this pilot study, the investigators aim to assess what the incidence of anterior vitrectomy is for each group, in order to better understand the sample size needed to assess whether there is a difference between these two groups. Secondarily, it will gather preliminary data on safety and refractive outcomes for patients undergoing these interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Los Angeles County + University of Southern California Medical Center (LAC+USC) who are 40 years or older with visually significant cataracts asking for surgical intervention.
* Cataract must be visually and clinically significant on examination as determined by the resident surgeon and the attending physician.

Exclusion Criteria:

* Age less than 40
* Visual acuity 20/30 or better with refraction in the study eye
* Any previous ocular surgery
* Patient request for monovision or for correction at near at the expense of distance
* Patient and physician decision to use an IOL implant other than monofocal IOL
* Corneal pathology (e.g. Fuch's dystrophy, corneal opacity or scar, corneal ectasia)
* Posterior or anterior capsular plaque
* Posterior polar cataract
* White cataract
* Subluxated lens, weak zonules, or phacodonesis
* Pseudoexfoliation syndrome
* Failure of preoperative pupillary dilatation (< 6 mm dilation)
* History of uveitis
* History of retinal detachment
* Untreated or active proliferative diabetic retinopathy
* Untreated or active diabetic macular edema
* Ocular diseases that may affect visual acuity or the operation (including and not limited to macular degeneration, retinitis pigmentosa, macular hole, advanced or end-stage glaucoma)
* Neurological or systemic diseases that may affect visual acuity or the safety of the operation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of anterior vitrectomy | 6 months
  Of all cases in each group, what percent results in any complication that needed conversion to anterior vitrectomy

SECONDARY OUTCOMES:
Incidence of dropped nucleus or intraocular lens (IOL) | 6 months
  Complication when the nucleus or implanted intraocular lens falls posteriorly
Incidence of posterior capsular tear | 6 months
  Complication where the posterior capsule is torn or ruptured
Incidence of anterior capsular tears or tags | 6 months
  Complication where the anterior capsule is torn or ruptured
Incidence of zonal injury | 6 months
  Complication where the cataractous nucleus or implanted IOL falls posteriorly.
Incidence of corneal injury | 6 months
  Complication when the cornea is injured during surgery
New onset macular edema | 6 months
  Presence of macular edema, by clinical evaluation or optical coherence tomography (OCT), which was not present before surgery
New onset ocular hypertension or glaucoma | 6 months
  Ocular hypertension or glaucoma, which was not present before surgery
Postoperative outcomes such as uncorrected and best corrected distance visual acuity | 6 months
  Measured by manifest refraction
Contrast sensitivity | 6 months
  Measured by Pelli-Robson Contrast Sensitivity Chart and the Contrast Sensitivity Testing (CSV-1000E)
Spherical equivalent | 6 months
  Calculated from the best corrected visual acuity
Corneal edema | 6 months
  Graded by the surgeon on a scale of 0 to 3 (none, mild, moderate, severe)
Central corneal thickness | 6 months
  Measured by pachymetry
Intraocular lens centration | 6 months
  Subjectively graded by the surgeon on a scale of 0 to 4 (poor, average, fair, excellent centration).
Educational gains of the resident surgeon | 6 months
  Done through surveys distributed to resident physicians throughout the course of the study